CLINICAL TRIAL: NCT07092917
Title: Surgical Outcomes and Complications of Posterior Spinal Fusion in Adolescent Idiopathic Scoliosis
Acronym: Scoliosis
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamad Sayed Mohamad, Assistant lecturer af neurosurgery, Assiut University
Other Study IDs: Scoliosis posterior
Record Dates: First submitted 2025-05-23; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Asses Radiological Efficacy of Posterior Approach Regarding Correction of Cobb Angle Post Operative . • Asses; Scoliosis Idiopathic Adolescent Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- posterior fusion surgery

SUMMARY:
Adolescent idiopathic scoliosis (AIS) is the most common form of scoliosis representing about 80-90% of all idiopathic scoliosis cases , characterized by lateral curvature of the spine of 10 degrees or more in children 10-18 years without underlaying cause .

AIS affects 1-3% of adolescents globally . More common in females with a ratio of 8;1 (1) The exact cause of AIS remain unknown ,however it's thought to be multi factorial may be due to genetic predisposition as it's often familial with multiple genetic loci impacting its pathogenesis heritability range between 30-60% (2) Bio mechanically the asymmetrical growth of the vertebrae and spinal loading may lead to curvature progression during rapid growth spurts Some studies suggest that asymmetrical loading of the spine can progress the deformity.

Multiple risk factors of progression have been detected: younger age at diagnosis , female sex ,higher initial Cobb angle and growth velocity (5) Severe scoliosis causes cosmetic concerns ,height reduction , reduced lung function and may progress to degenerative changes in adulthood (6) Treatment options for AIS include observation , bracing and surgery for curves more than 40 degree Cobb angle (7) Surgical correction has been a controversy for many years depending on the severity of the curve , the facility , surgeons preference and available instrumentation.

Anterior surgery became popular due to some advantage over posterior surgery as direct derotation of the spine ,removal of the disc ,over correction of the apex over short construct but some results from that correction is production of hyper kyphosis which can cause pulmonary problems ,anterior surgery carry high risk of pseudoarthrosis ,increase motion stress distal to corrected levels causing adjacent level disease Anterior surgery also requires high degree of flexibility in curve otherwise it is not applicable .

With advancing technique in posterior surgery and multiple training ,posterior surgery have been widely employed in correction of AIS with the same or even better results in severe cases As there is minimal affection in pulmonary function also it provides correction of Sagittal balance. (8)

DETAILED DESCRIPTION:
Adolescent idiopathic scoliosis (AIS) is the most common form of scoliosis representing about 80-90% of all idiopathic scoliosis cases , characterized by lateral curvature of the spine of 10 degrees or more in children 10-18 years without underlaying cause .

AIS affects 1-3% of adolescents globally . More common in females with a ratio of 8;1 (1) The exact cause of AIS remain unknown ,however it's thought to be multi factorial may be due to genetic predisposition as it's often familial with multiple genetic loci impacting its pathogenesis heritability range between 30-60% (2) Bio mechanically the asymmetrical growth of the vertebrae and spinal loading may lead to curvature progression during rapid growth spurts Some studies suggest that asymmetrical loading of the spine can progress the deformity.

Multiple risk factors of progression have been detected: younger age at diagnosis , female sex ,higher initial Cobb angle and growth velocity (5) Severe scoliosis causes cosmetic concerns ,height reduction , reduced lung function and may progress to degenerative changes in adulthood (6) Treatment options for AIS include observation , bracing and surgery for curves more than 40 degree Cobb angle (7) Surgical correction has been a controversy for many years depending on the severity of the curve , the facility , surgeons preference and available instrumentation.

Anterior surgery became popular due to some advantage over posterior surgery as direct derotation of the spine ,removal of the disc ,over correction of the apex over short construct but some results from that correction is production of hyper kyphosis which can cause pulmonary problems ,anterior surgery carry high risk of pseudoarthrosis ,increase motion stress distal to corrected levels causing adjacent level disease Anterior surgery also requires high degree of flexibility in curve otherwise it is not applicable .

With advancing technique in posterior surgery and multiple training ,posterior surgery have been widely employed in correction of AIS with the same or even better results in severe cases As there is minimal affection in pulmonary function also it provides correction of Sagittal balance. (8)

ELIGIBILITY:
Inclusion Criteria:

* • Male and female Adolescents aged 10 to 18 years diagnosed with AIS

  * Patients with Risser sign 4 and 5 indicating maturity of the skeletal system
  * Patents with lenke classification system 2,3,4
  * Curvature between 40 and 70 degrees Cobb angle indicating moderate to severe scoliosis suitable for surgical correction
  * Candidates for surgical intervention due to rapid progression of deformity more than 5 degrees per year ,functional limitations

Exclusion Criteria:

* • Congenital or neuromuscular scoliosis

  * Pre operative restrictive lung function
  * Previous spinal surgery
  * Severe co morbidities preventing surgical intervention .

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Inclusion Criteria:
  * • Male and female Adolescents aged 10 to 18 years diagnosed with AIS
    * Patients with Risser sign 4 and 5 indicating maturity of the skeletal system
    * Patents with lenke classification system 2,3,4
    * Curvature between 40 and 70 degrees Cobb angle indicating moderate to severe scoliosis suitable for surgical correction
    * Candidates for surgical intervention due to rapid progression of deformity more than 5 degrees per year ,functional limitations
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2027-08-15 (Estimated); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
clinical evaluation of the patients height thoracic symmetry rib humb | 2 years
  comparison between peoperative and post operative measures of shoulder height , waist symmetry by measures of pelvic tilt .
Cobb angle | 2 years
  Comparison between pre and post op Cobb angle
functional outcome of patients satisfaction after surgery | 2 years
  measuring the functional outcome post surgery regarding pain and disability using SRS-22 score , VAS score for pain and Oswestry disability index

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university hospitals, Asyut, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: No